# Note to File:

# Statistical Analysis for the VAC 049 Abbreviated CSR

# Study Title:

A Phase 1 Randomized, Double-Blinded, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability and Immunogenicity of Live Attenuated, Oral Shigella WRSS1 Vaccine in Bangladeshi Toddlers (12 to 24 months old)

Version 1.0

04 October 2018

Prepared and distributed by:

The Emmes Corporation

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

**Study Title:** A Phase 1 Randomized, Double-Blinded, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability and Immunogenicity of Live Attenuated, Oral Shigella WRSS1 Vaccine in Bangladeshi Toddlers (12 to 24 months old).

| Trial Number Code: | Protocol: VAC 049 |
|---|---|
| Development Phase: | Phase I |
| Investigational Products: | Live attenuated S. sonnei WRSS1 |
| Sponsor: | PATH Vaccine Solutions |
| Principal Investigator | Rubhana Raqib, PhD Infectious Diseases Division, icddr,b 68 Shaheed Tajuddin Ahmed Sarani, Mohakhali, Dhaka-1212, Bangladesh |
| Co-Principal Investigator/ Study Physician: | K. Zaman, MD PhD Infectious Diseases Division, icddr,b 68 Shaheed Tajuddin Ahmed Sarani, Mohakhali, Dhaka-1212, Bangladesh |
| Clinical Trial Operational Oversight | PATH 2201 Westlake Avenue, Suite 200 Seattle, WA 98121 USA |
| Biostatistician: | Len Dally The Emmes Corporation 401 North Washington Street, Suite 700 Rockville, MD 20850 USA |
| Clinical Trial Initiation Date: | 23 February 2017 |
| Clinical Trial Completion Date: | 10 January 2018 |
| Date of Clinical Study Report: | 04 April 2018 |
| Version of Clinical Study Report: | v 1.0 |

#### SIGNATURE PAGE

STUDY TITLE:

A Phase 1 Randomized, Double-Blinded, Placebo-Controlled, Dose-Escalation Study to Assess the Safety, Tolerability and Immunogenicity of Live Attenuated, Oral Shigella WRSS1 Vaccine in Bangladeshi Toddlers (12 to 24 months old)

PROTOCOL NUMBER: VAC 049

PATH Medical Officer: Tushar Tewari, MD

The Emmes Corporation Statistician: Len Dally, MS

Signed:

## **Table of Contents**

| atistical A | nalysis for the VAC 049 Abbreviated CSR | 1 |
|---|---|---|
| SIGNATU | IRE PAGE | 3 |
| Introduc | tion | 7 |
| Purpose | of the Analysis | 7 |
| - | • | |
| 2.2 Sec | condary Study Hypotheses | 7 |
| Study O | bjectives | 7 |
| 3.2 Sec | condary Study Objectives | 8 |
| 3.3 Exp | oloratory Objectives | 8 |
| Study D | esign | 8 |
| Study P | rocedures/Evaluations | 9 |
| Assessn | nent of Safety | 9 |
| Sample | Size Calculation and Outcome Primary and Secondary Variables | 9 |
| 7.1 Sar | nple Size | 9 |
| 7.2 Fina | al Data Analysis | 9 |
| 7.2.1 | Analysis Populations | 9 |
| 7.2.2 | General Analytic Plan | 10 |
| 7.2.3 | Safety Analysis | 10 |
| 7.2.4 | Immunogenicity Analysis: | 11 |
| Referen | ces | 11 |
| Appendi | x I: Table Shells | 12 |
| | SIGNATU Introduct Purpose 2.1 Prir 2.2 Sec Study O 3.1 Prir 3.2 Sec 3.3 Exp Study D Study Pr Assessn Sample 7.1 San 7.2 Fina 7.2.1 7.2.2 7.2.3 7.2.4 Referen | 2.2 Secondary Study Hypotheses Study Objectives 3.1 Primary Study Objective |

# **List of Tables**

| Figure 1. CONSORT Diagram | 12 |
|---|---|
| Table 7.1 Summary of Participant Disposition – All Participants | 13 |
| Table 7.2 Summary of Analysis Populations | 13 |
| Table 7.3 Summary of Demographic Characteristics – Safety Population | |
| Table 7.4 Summary of Medical History at Screening | 15 |
| Table 7.5 Summary of Abnormal Physical Examination Results at Screening | 16 |
| Table 7.6 Summary of Protocol Deviation | |
| | 18 |
| Table 8.2.1 Maximum Severity of Any Systemic Reactogenicity by Vaccination in Cohort C1 - Safety Population | 19 |
| Table 8.2.2 Maximum Severity of Fever by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.3 Maximum Severity of Decreased Appetite by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.4 Maximum Severity of Irritability by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.5 Maximum Severity of Decreased Activity by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.6 Maximum Severity of Any Intestinal Reactogenicity by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.7 Maximum Severity of Abdominal Pain by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.8 Maximum Severity of Nausea by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.9 Maximum Severity of Vomiting by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.10 Maximum Severity of Loose Stool by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.11 Maximum Severity of Diarrhea by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.12 Maximum Severity of Dysentery by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.13 Maximum Severity of Bloating by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.14 Maximum Severity of Excess Flatulence by Vaccination in Cohort C1 - Safety Population. | |
| Table 8.2.15 Maximum Severity of Constipation by Vaccination in Cohort C1 - Safety Population | |
| Table 8.2.16 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Any Vaccination in | 21 |
| Table 8.2.17 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Vaccination 1 in | 22 |
| Table 8.2.18 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Vaccination 2 in | |
| | 22 |
| Table 8.2.19 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Vaccination 3 in | |
| Cohort C1 - Safety Population | 22 |
| Table 8.2.20 Intestinal Reactogenicity of Grade 2 or Greater Severity by Day Post Any Vaccination in | |
| | 23 |
| Table 8.2.21 Intestinal Reactogenicity of Grade 2 or Greater by Day Post Vaccination 1 in Cohort C1 - | <u> </u> |
| | 24 |
| | 24 |
| Table 8.2.23 Intestinal Reactogenicity of Grade 2 or Greater by Day Post Vaccination 3 in Cohort C1 - Safety Population | 24 |
| Table 8.2.24 Maximum Severity per Participant of Unsolicited Adverse Events Occurring within | |
| 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC and PT - Safety Population 2 | 25 |
| Table 8.2.25 Maximum Severity per Participant of Unsolicited Adverse Events Related to Study Product Occurring Within 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC | |
| and PT - Safety Population | 26 |
| Table 8.2.26 Maximum Severity per Participant of Unsolicited Serious Adverse Events(SAE) Occurring Within 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC and PT - Safety | |
| Population | 26 |
| Table 8.2.27 Maximum Severity per Participant of Unsolicited Serious Adverse Events(SAE) Related | |
| to Study Product Occurring Within 28 Days After Any Vaccination in Cohort C1, by | |
| MedDRA SOC and PT - Safety Population | 26 |
| Table 8.2.28 Maximum Severity per Participant of Unsolicited Adverse Events Occurring Within 28 Days After Vaccination 1 in Cohort C1, by MedDRA SOC and PT - Safety Population | 26 |

| Table 8.2.29 Maximum Severity per Participant of Unsolicited Adverse Events Occurring Within 28 Days After Vaccination 2 in Cohort C1, by MedDRA SOC and PT - Safety Population | . 26 |
|---|---|
| Table 8.2.30 Maximum Severity per Participant of Unsolicited Adverse Events Occurring Within 28 | |
| Days After Vaccination 3 in Cohort C1, by MedDRA SOC and PT - Safety Population | . 26 |
| Table 8.2.31 Maximum Severity per Participant of Unsolicited Adverse Events Related to Study | |
| Product Occurring Within 28 Days After Vaccination 1 in Cohort C1, by MedDRA SOC and | |
| PT - Safety Population | . 26 |
| Table 8.2.32 Maximum Severity per Participant of Unsolicited Adverse Events Related to Study | _ |
| Product Occurring Within 28 Days After Vaccination 2 in Cohort C1, by MedDRA SOC and | |
| PT - Safety Population | . 26 |
| Table 8.2.33 Maximum Severity per Participant of Unsolicited Adverse Events Related to Study | |
| Product Occurring Within 28 Days After Vaccination 3 in Cohort C1, by MedDRA SOC and | |
| PT - Safety Population | . 26 |
| Table 8.2.34 Overall Incidence of Unsolicited Serious Adverse Events Within 28 Days After | |
| Vaccination, by Vaccination in Cohort C1 - Safety Population | . 27 |
| Table 8.3.1 Listing of Unsolicited Non-Serious Adverse Events of Grade 2 or Greater Severity in | |
| Participants in Cohort C1 - Safety Population | . 28 |
| Table 8.3.2 Listing of Unsolicited Serious Adverse Events in Participants in Cohort C1 - Safety | |
| Population | . 28 |
| Table 8.4.1 Listing of all Hematology and Biochemistry Results in Participants in Cohort C1 with any | |
| Grade 2 or Greater Severity - Safety Population | |
| Table 8.5.1 Listing of all Physical Examination and Vital Signs Values in Participants in Cohort C1 with | |
| Any Abnormality Findings - Safety Population | |
| Table 10.2.1 IgA Antibodies in ALS, Descriptive Statistics - Per Protocol Population | |
| Table 10.2.2 IgG Antibodies in ALS, Descriptive Statistics - Per Protocol Population | |
| Table 10.2.3 IgM Antibodies in ALS, Descriptive Statistics - Per Protocol Population | |
| Table 10.2.4 Fold-Rise from Baseline in IgA Antibodies in ALS – Per-Protocol Population | |
| Table 10.2.5 Fold-Rise from Baseline in IgG Antibodies in ALS – Per-Protocol Population | |
| Table 10.2.6 Fold-Rise from Baseline in IgM Antibodies in ALS – Per-Protocol Population | . 32 |
| Table 10.2.7 4-Fold Rise <sup>1</sup> in IgA Antibodies in ALS Proportion of Participants with at Least a 4-Fold | |
| Rise from Baseline – Per-Protocol Population | . 33 |
| Table 10.2.8 4-Fold Rise in IgG Antibodies in ALS Proportion of Participants with at Least a 4-Fold | |
| Rise from Baseline – Per-Protocol Population | . 34 |
| Table 10.2.9 4-Fold Rise in IgM Antibodies in ALS Proportion of Participants with at Least a 4-Fold | |
| Rise from Baseline – Per-Protocol Population | |
| Table 10.2.10 - Table 10.2.12 Replicate Table 10.2.1-10.2.3 for IgA, IgG and IgM Antibodies in Serum | . 34 |
| Table 10.2.13 - Table 10.2.15 Replicate Table 10.2.4-10.2.6 for IgA, IgG and IgM Antibodies in Serum | . 34 |
| Table 10.2.16 - Table 10.2.18 Replicate Table 10.2.7-10.2.9 for IgA, IgG and IgM Antibodies in Serum | . 34 |
| Table 10.2.19 Replicate Table 10.2.1 for IgA Antibodies in Stool – Per Protocol Population, include | |
| extra visits (Days 28, 56 and 84) | . 34 |
| Table 10.2.20 Replicate Table 10.2.4 for IgA Antibodies in Stool – Per Protocol Population, include | |
| extra visits (Days 28, 56 and 84) | . 34 |
| Table 10.2.21 Replicate Table 10.2.7 for IgA Antibodies in Stool – Per Protocol Population, include | |
| extra visits (Days 28, 56 and 84) | . 34 |
| Table 10.2.22 Proportion of Participants with WRSS1 Shedding at Any Time after Vaccination – | |
| Per-Protocol Population | . 34 |
| 1. Listing of Participants Withdrawn | |
| 2. Listing of Demographic and Other Baseline Characteristics | |
| 3. Listing of Medical History | |
| 4. Listing of Physical Examination Results | . 35 |
| 5. Listing of Protocol Deviations | |
| 6. Listing of Participant Vaccinations | |

## 1 Introduction

This is a note to file generated to provide a detailed summary of analysis conducted for VAC 049 abbreviated clinical study report. This was a single site, Phase 1, double-blind, randomized, placebo-controlled, dose-escalation study in toddlers (12-24 months old). The study was intended to enroll approximately 64 toddlers (12-24 months old) in 4 groups of 16, to receive three doses of 3x10³, 3x10⁴, 3x10⁵ or 3x10⁶ CFU WRSS1 vaccine or placebo (sterile saline solution). However, only the 16 participants in Cohort C1 (3x10³ WRSS1(n=12) or placebo (n=4) with 3:1 randomization ratio) were enrolled and vaccinated as enrollment was terminated after Cohort C1 because the funder, the Bill and Melinda Gates Foundation (BMGF), made significant changes to the PATH Enteric Vaccine Initiative (EVI) portfolio and elected to discontinue support of the study, prior to enrollment of three higher-dose cohorts. Notification of study termination was sent to the FDA on October 4, 2017 as part of SN0015. As the study was terminated prematurely and prior to the development of a formal Statistical Analysis Plan (SAP), table shells were developed based on the statistical analysis sections in the study protocol, prior to completing the final analyses. In lieu of a full SAP, this note to file provides additional analysis details along with the previously-approved table shells for study documentation and archiving purposes.

# 2 Purpose of the Analysis

### 2.1 Primary Study Hypothesis

 Orally administered WRSS1 would be safe and tolerable in toddler recipients and would cause no major side effects in vaccinated participants.

### 2.2 Secondary Study Hypotheses

- WRSS1 was to generate a positive (4-fold rise in serum/plasma) immune response detectable in one or more assays in at least 50% of vaccinees.
- WRSS1 was to be able to replicate in the intestine as determined by fecal shedding.

# 3 Study Objectives

## 3.1 Primary Study Objective

To evaluate the safety and clinical tolerance of WRSS1 in Bangladeshi toddlers (12-24 months old) by monitoring the occurrence and severity of clinical signs and symptoms after administration of three vaccine doses. All the analyses were to be performed by dose groups.

Safety was to be assessed by analyses of the following primary endpoints (events), where the unit of analysis in each case will be the proportion of participants with at least one event:

- any solicited reactogenicity
- any unsolicited AEs
- any SAEs
- unsolicited AEs and SAEs judged as having a reasonable possibility that the study product caused the event

### 3.2 Secondary Study Objectives

- To examine the immunogenicity of WRSS1.
- To assess the ability to replicate and duration of fecal shedding of WRSS1 following ingestion.

The secondary immunogenicity endpoints were chosen to further assess the mucosal and systemic immunogenicity. This was done by assessing:

- Frequency and magnitude of antigen specific serum IgG, IgA and IgM antibody titers to S. sonnei LPS, and S. sonnei Invaplex antigens after administration of one or three vaccine doses
- Frequency and magnitude of antigen-specific fecal IgA antibody titer to *S. sonnei* LPS and *S. sonnei* Invaplex antigens after administration of one or three vaccine doses
- Frequency and magnitude of antigen (LPS and Invaplex)-specific IgG, IgA, and IgM antibody titers in lymphocyte supernatant (ALS) to *S. sonnei* LPS and Invaplex antigens.

Finally, fecal shedding of vaccine was measured by the frequency and duration of detectable fecal presence of WRSS1 by culture and PCR.

#### 3.3 Exploratory Objectives

To evaluate serum bactericidal activity and cytokine profile against WRSS1 in toddlers before and after vaccination.

# 4 Study Design

This was a single site, Phase 1, double-blind, randomized, placebo-controlled, dose-escalation study in toddlers (12-24 months old). The study was intended to enroll approximately 64 toddlers (12-24 months old) in 4 groups of 16, to receive three doses of  $3x10^3$ ,  $3x10^4$ ,  $3x10^5$  or  $3x10^6$  CFU WRSS1 vaccine or placebo (sterile saline solution). However, only the 16 participants in Cohort C1 ( $3x10^3$  WRSS1(n=12) or placebo (n=4) with 3:1 randomization ratio) were enrolled and vaccinated as enrollment was terminated after Cohort C1 because the funder, the Bill and Melinda Gates Foundation (BMGF), made significant changes to the PATH Enteric Vaccine Initiative (EVI) portfolio and elected to discontinue support of the study, prior to enrollment of three higher-dose cohorts. Notification of study termination was sent to the FDA on October 4, 2017 as part of SN0015.

For full study details, please refer to Section 4 (Research Design and Methods) of the VAC 049 study protocol.

# 5 Study Procedures/Evaluations

Please refer to the following sub-sections from Sections 7 (Study Procedures/Evaluations), 8 (Study Schedule), and the Appendix I (Time and Event Schedule) of the VAC 049 study protocol:

- 7.1 Clinical Definitions
- 7.2 Concomitant Medication/Treatments
- 7.3 Laboratory Evaluations
- 8.1 Screening, Days -30 to -9 (Visit 01)
- 8.2 Day of First Vaccination (Visit 02)
- 8.3 Inpatient Period (Visit 03)
- 8.4 Discharge (Visit 03)
- 8.5 Outpatient Visits
- 8.6 Early Termination

# 6 Assessment of Safety

Please refer to the following sub-sections from Section 10 (Assessment of Safety) of the VAC 049 study protocol:

- 10.1.1 Adverse Event Definitions
- 10.1.2 Reactogenicity
- 10.1.3 Guidelines for Determine Causality of an Adverse Event
- 10.2 Safety Oversight Data Safety Monitoring Board (DSMB)

# 7 Sample Size Calculation and Outcome Primary and Secondary Variables

#### 7.1 Sample Size

Please refer to the following sub-sections from Section 12 (Sample size Calculation and Outcome Primary and Secondary Variables) of the VAC 049 study protocol:

- 12.1 Introduction
- 12.2 Sample Size

#### 7.2 Final Data Analysis

Only Cohort C1 was enrolled and vaccinated, so all data analyses were limited to Cohort C1. All decisions about data analysis were made prior to database freeze and the final analyses were conducted after database freeze.

#### 7.2.1 Analysis Populations

**Safety Population:** all enrolled participants who were randomized to either WRSS1 or Placebo and were vaccinated. This population was used in the analysis of all safety, study population, demographic & baseline characteristics data.

**Per-Protocol Population**: all randomized participants who received all three vaccinations and provided any immunology data through Day 84. This population was defined and interpreted based on the criteria in Section 12.3.2 of the study protocol, which stated that the analysis of

immunogenicity will include all participants who provide specimens through Day 84. This population was used in the analysis of all immunogenicity data.

The analysis populations were defined during blinded table shell preparation in collaboration between the sponsor and the CRO before final database lock and before breaking the blind.

#### 7.2.2 General Analytic Plan

- I. In this trial, only Cohort C1 was enrolled. Subjects were administered 3 doses of vaccine (3 X 10<sup>3</sup> CFU) or placebo, per randomized allocation, on Days 0, 28, and 56.
- II. Shells for table, listing and figures are presented in Appendix I of this Note to File.
- III. When the use of descriptive statistics to assess group characteristics was required, the following methods were to be used: for categorical variables, the number and percent in each category; for continuous variables, mean (with standard deviation), median, geometric mean and range (minimum, maximum).
- IV. For statistical comparison between arms, the Chi-square test (if all expected frequencies in a table were >5) or Fisher's exact test for categorical variables, and Student's *t*-test for continuous variables were to be utilized. The Clopper-Pearson exact two-sided 95% Cl's were to be presented for within group proportion estimates, while the *t*-distribution was to be utilized to estimate the two-sided 95% Cl's of within group estimates of geometric mean and between-group geometric mean fold-rise.
- V. Demographic, baseline, and other study population data were to be summarized descriptively. These tables include participant disposition, analysis populations, demographic characteristics, medical history, abnormal physical examination and protocol deviations (Tables 7.1-7.6). Listings corresponding to the above descriptive summary tables were also to be generated.
- VI. Due to the exploratory nature of the study, no adjustment was to be made for multiple testing. No imputation of missing data was to be performed as the complete samples among those in the analysis populations at each time point were to be analyzed.
- VII. All analyses were to be unadjusted for potential covariates.

#### 7.2.3 Safety Analysis

All visits after the participants had been exposed to the study product were to be included in the primary analysis of safety. To assess safety, the number and the percentages of participants experiencing at least one AE, and the number and percentage of participants experiencing each specific AE was to be tabulated according to maximum severity and relationship by study arm by both, overall and after each vaccination.

Analysis of safety data includes Tables 8.2.1 - 8.2.34, 8.3.1 - 8.5.1 Note that tables were numbered as Tables 9.2.1 - 9.2.34, 9.3.1 - 9.5.1 in CSR. The following describes the planned analysis for safety data:

- Descriptive summary and statistical comparison (WRSS1 vs Placebo) of solicited systemic reactogenicity
- Descriptive summary and statistical comparison (WRSS1 vs Placebo) of solicited intestinal reactogenicity
- Descriptive summary of unsolicited adverse event by MedDRA SOC and PT
- Listing of adverse events, serious adverse events, death (including narrative)
- Listing of Hematology and Biochemistry

#### 7.2.4 Immunogenicity Analysis:

The magnitude of IgA, IgG and IgM ALS, and serum measures were to be evaluated on Days 0, 7, 35 and 63, while the magnitude of IgA fecal measures were to be evaluated on Days 0, 7, 28, 35, 56, 63, and 84. A fold rise response was to be defined as a 4-fold increase in titer value at a post-baseline visit when compared to the baseline visit (Day 0). The response rate was summarized for each post-baseline time point using the number and percent, and including two-sided 95% exact confidence intervals for the rate. Immune measures were to be measured against *S. sonnei* LPS and Invaplex antigens and hence, analyzed separately.

Analysis of immunology data includes Table 10.2.1 – 10.2.22. Note that tables were numbered as Tables 11.2.1 – 11.2.21 in the CSR and Table 10.2.22 was not produced since no data were available. The following describes the planned analysis for immunology data:

- Descriptive summary of IgA, IgG, and IgM in ALS and Serum
- Descriptive summary and statistical comparison (WRSS1 vs Placebo) of fold-rise from baseline, based on the ratio of follow-up to baseline titers, in IgA, IgG, and IgM in ALS and Serum
- Descriptive summary and statistical comparison (WRSS1 vs Placebo) of 4-fold rise, based on the ratio of follow-up to baseline titers, in IgA, IgG, and IgM in ALS and Serum.
- Descriptive summary of IgA, in Stool
- Descriptive summary and statistical comparison (WRSS1 vs Placebo) of fold-rise, based on the ratio of follow-up to baseline titers, from baseline in IgA in stool.
- Descriptive summary and statistical comparison (WRSS1 vs Placebo) of 4-fold rise, based on the ratio of follow-up to baseline titers in IgA in stool.
- Proportion of Participants with WRSS1 Shedding at any time after vaccination

# 8 References

- 1. Study Protocol: PR16023\_VAC 049\_V4\_14Feb2017
- 2. Study CSR: VAC049 Abbreviated-CSR 04Apr2018 v1.0

# 9 Appendix I: Table Shells

Assessed for Eligibility Screened but not enrolled (n=xx)  $(n-\infty)$  Withdrew consent (n=xx) Did not meet eligibility criteria (n=xx) Accrual goals already met (n=xx). Falled continued eligibility on Day 0 (n=xx). Randomized (n=xx) Cohort C1 Cohort C1 Cohorts C2, C3 & C4 (3 x 10° CFU WRSS1) Study did not (Placebo) Received 1" dose at Received 1st dose at progress to Cohort C2, C3 and C4 Day 0 (n=xx)Day 0 (n=xx) Received 2nd dose at Received 2nd dose at Day 28 (n=xx) Day 28 (n=xx) Received 3rd dose at Received 3rd dose at Day 56 (n=xx) Day 56 (n-xx) Completed Completed follow-up follow-up (n-xx)(n-xx)Analyzed: Analyzed Vaccine (n=xx) Vaccine (n=xx) Placebo (n=x) Placebo (n=x).

Figure 1. CONSORT Diagram

Table 7.1 Summary of Participant Disposition - All Participants

| | Cohort C1 | | |
|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
| Screened | N/A | N/A | |
| Enrolled | N/A | N/A | |
| Randomized | | | |
| Participants completed the study | | | |
| Yes | | | |
| No | | | |
| If no, reason for premature termination | | | |
| Serious Adverse Event (other than death) | | | |
| Adverse Event, other than SAE | | | |
| Lost for Follow-up | | | |
| Non-Compliance/Protocol Deviation | | | |
| Voluntary Withdrawal by Participants/Parent | | | |
| Withdrawal by Investigator | | | |
| Termination of Site or Study by Sponsor | | | |
| Death | | | |
| Enrolled but not Vaccinated/Treated | | | |
| Others | | | |

N= Number of participants screened and, n= Number of participants as per row description.

N/A: Not Applicable.

Source: Listing 1. Listing of Participants Withdrawal

**Table 7.2 Summary of Analysis Populations** 

| | | Cohort C1 | |
|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
| Safety Population | | | |
| Per-Protocol Population | | | |

N=Number of participants randomized and, n= is number of participants as per row description.

Percentages are calculated based on all screened participants while disposition details are calculated based on all randomized participants.

Denominator of the percentage is the number of randomized participants in the respective groups except for the 'Screened' and 'Enrolled' row.

**Table 7.3 Summary of Demographic Characteristics – Safety Population** 

| | Cohort C1 | | |
|---|---|---|---|
| Characteristics | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX) | Placebo<br>(N=XX) | Total<br>(N=XX) |
| Gender, n (%) | · | | |
| Female | | | |
| Male | | | |
| Age (Years) | <u>.</u> | | |
| n | | | |
| Mean (STD) | | | |
| Median (Min, Max) | | | |
| Race, n (%) | - | | |
| Black | | | |
| White | | | |
| Asian | | | |
| Height (cm) | • | | |
| n | | | |
| Mean (STD) | | | |
| Median (Min, Max) | | | |
| Weight (Kg) | | | |
| n | | | |
| Mean (STD) | | | |
| Median (Min, Max) | | | |

N= Number of participants in the Safety Population and, n= Number of participants with non-missing data.

Denominator of the percentage is the number of non-missing participants in Safety Population within the respective groups.

Source: Listing 2. Listing of Demographic and other Baseline Characteristics

**Table 7.4 Summary of Medical History at Screening** 

| | | Cohort C1 | |
|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
| HEENT | | | |
| HEENT-Head | | | |
| HEENT-Eyes | | | |
| HEENT-Ears | | | |
| HEENT-Nose | | | |
| HEENT-Throat/Mouth | | | |
| Cardiovascular | | | |
| Cardiovascular-Heart/Veins or Arteries | | | |
| Respiratory | | | |
| Gastrointestinal | | | |
| Gastrointestinal-Stomach | | | |
| Gastrointestinal-Intestines | | | |
| Hepatobiliary/Pancreas | | | |
| Liver/Pancreas | | | |
| Gall bladder | | | |
| Urologic | | | |
| Neurologic | | | |
| Autoimmune Disease | | | |
| Previous Vaccination | | | |
| No | | | |
| Yes | | | |
| Polio | | | |
| BCG | | | |
| Rotavirus | | | |
| Others | | | |

N= Number of participants in the Safety Population; n= Number of participants as per row description.

Denominator of the percentage is the number of non-missing participants in Safety Population within the respective groups. Source: Listing 3. Listing of Medical History

Table 7.5 Summary of Abnormal Physical Examination Results at Screening

| | Cohort C1 | | |
|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX) | Placebo<br>(N=X) | Total<br>(N=X) |
| Area/System | n (%) | n (%) | n (%) |
| HEENT | | | |
| Skin | | | |
| Cardiovascular (heart) | | | |
| Respiratory (lung) | | | |
| Abdomen | | | |
| Musculoskeletal | | | |
| Neurological | | | |
| Lymph Nodes | | | |
| Other | | | |

N= Number of participants in the Safety Population and n= Number of participants as per row description.

Denominator of the percentage is the number of participants in Safety Population within the respective groups.

Source: Listing 4. Listing of Physical Examination Results

**Table 7.6 Summary of Protocol Deviation** 

| | Cohort C1 | | |
|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX)<br>n (%) | Placebo<br>(N=XX)<br>n (%) | Total<br>(N=XX)<br>n (%) |
| Participant is Protocol Deviation | | | |
| Yes | | | |
| No | | | |
| If Yes, reason for protocol deviation | | | |
| Participant illness | | | |
| Participants unable to comply | | | |
| Participant/ parent refusal | | | |
| Clinic Error | | | |
| Pharmacy Error | | | |
| Laboratory Error | | | |
| Investigator/Study Decision | | | |
| Others | | | |
| Deviation resulted in an AE | | | |
| Deviation resulted in participant termination of study follow up | | | |
| Deviation affects or potentially affect, product stability | | | |
| Deviation Category | | | |
| Eligibility/enrollment | | | |
| Product administration schedule | | | |
| Follow up visit schedule | | | |
| Protocol Procedure/assessment | | | |
| Protocol administration | | | |
| Blinding policy/procedure | | | |
| Deviation met IRB reporting requirements | | | |

N= Number of participants in the Safety Population and n= Number of participants as per row description.

Denominator of the percentage is the number of participants in Safety Population within the respective groups. **Source**: Listing 5. Listing of Protocol Deviations

**Table 8.1 Summary of Participant Vaccinations** 

| | Cohort C1 | | |
|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX) | Placebo<br>(N=X) | Total<br>(N=X) |
| Vaccination | n (%) | n (%) | n (%) |
| Received Vaccination #1 | | | |
| Received Vaccination #2 | | | |
| Received Vaccination #3 | | | |
| Received All Vaccinations | | | |

N= Number of participants in the Safety Population and n= Number of participants as per row description.

Denominator of the percentage is the number of participants in Safety Population within the respective groups.

Source: Listing 6. Listing of Participant Vaccinations

Table 8.2.1 Maximum Severity of Any Systemic Reactogenicity by Vaccination in Cohort C1 - Safety Population

| | | Cohort C1 | | | |
|---|---|---|---|---|---|
| | (3 x 10 | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX) | | cebo<br>=X) | P-value<br>(Vaccine vs |
| | x/n (%) | 95% CI | x/n (%) | 95% CI | Placebo) |
| Maximum Overall | | | | | |
| Mild | | | | | 0.xxx <sup>1</sup> |
| Moderate | | | | | |
| Severe | | | | | |
| Potential Life Threatening | | | | | |
| Any Severity | | | | | $0.xxx^2$ |
| Post Vaccination 1 | | | | | |
| Mild | | | | | 0.xxx <sup>1</sup> |
| Moderate | | | | | - |
| Severe | | | | | |
| Potential Life Threatening | | | | | • 2 |
| Any Severity | | | | | $0.xxx^2$ |
| Post Vaccination 2 | | | | | |
| Mild | | | | | 0.xxx <sup>1</sup> |
| Moderate | | | | | |
| Severe | | | | | |
| Potential Life Threatening | | | | | 2 2 |
| Any Severity | | | | | 0.xxx <sup>2</sup> |
| Post Vaccination 3 | | | | | |
| Mild | | | | | 0.xxx <sup>1</sup> |
| Moderate | | | | | |
| Severe | | | | | |
| Potential Life Threatening | | | | | 2 3 |
| Any Severity | | | | | $0.xxx^2$ |

N=Number of participants in the Safety Population.

Grades are based on maximum severity per participant.

Cells show frequency (x) and percent of participants with events.

n = number of participants that received vaccination.

CI = Exact 95% Confidence Interval for the proportion.

For Fever: Mild:  $\geq$ 100.4°F (38°C), Moderate: >101.1°F (38.5°C), Severe: >102.0°F (39°C), Potentially Life-Threatening>104.0°F (40°C)

Note: tables for any intestinal reactogenicity event and other individual reactogenicity events (8.2.2 - 8.2.15) will have similar shells.

<sup>&</sup>lt;sup>1</sup>Chi-square or Fisher's exact 2-tailed test if conditions for chi-square test are not satisfied.

<sup>&</sup>lt;sup>2</sup>Chi-square or Fisher's exact 1-tailed test of more events in the WRSS1 arms than in the placebo arm.

- Table 8.2.2 Maximum Severity of Fever by Vaccination in Cohort C1
   Safety Population
- Table 8.2.3 Maximum Severity of Decreased Appetite by Vaccination in Cohort C1
   Safety Population
- Table 8.2.4 Maximum Severity of Irritability by Vaccination in Cohort C1
   Safety Population
- Table 8.2.5 Maximum Severity of Decreased Activity by Vaccination in Cohort C1
   Safety Population
- Table 8.2.6 Maximum Severity of Any Intestinal Reactogenicity by Vaccination in Cohort C1 Safety Population
- Table 8.2.7 Maximum Severity of Abdominal Pain by Vaccination in Cohort C1
   Safety Population
- Table 8.2.8 Maximum Severity of Nausea by Vaccination in Cohort C1 Safety Population
- Table 8.2.9 Maximum Severity of Vomiting by Vaccination in Cohort C1 Safety Population
- Table 8.2.10 Maximum Severity of Loose Stool by Vaccination in Cohort C1
   Safety Population
- Table 8.2.11 Maximum Severity of Diarrhea by Vaccination in Cohort C1
   Safety Population
- Table 8.2.12 Maximum Severity of Dysentery by Vaccination in Cohort C1
   Safety Population
- Table 8.2.13 Maximum Severity of Bloating by Vaccination in Cohort C1
   Safety Population
- Table 8.2.14 Maximum Severity of Excess Flatulence by Vaccination in Cohort C1
   Safety Population
- Table 8.2.15 Maximum Severity of Constipation by Vaccination in Cohort C1
   Safety Population

Table 8.2.16 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post
Any Vaccination in Cohort C1 - Safety Population

| | | Coh | ort C1 | |
|---|---|---|---|---|
| | (3 x 1 | RSS1<br>I0³ CFU)<br>I=XX) | | ıcebo<br>√=X) |
| | x/n (%) | 95% CI | x/n (%) | 95% CI |
| Maximum Overall | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Fever | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Decreased Appetite | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Irritability | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Decreased Activity | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |

N=Number of participants in the Safety Population.

Cells show frequency (x) and percent of participants with events. n represent number of participants that received vaccination.

CI = Exact 95% Confidence Interval for the proportion.

For Fever: Mild: ≥100.4°F (38°C), Moderate: >101.1°F (38.5°C), Severe: >102.0°F (39°C), Potentially Life-Threatening>104.0°F (40°C)

- Table 8.2.17 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Vaccination 1 in Cohort C1 Safety Population
- Table 8.2.18 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Vaccination 2 in Cohort C1 Safety Population
- Table 8.2.19 Systemic Reactogenicity of Grade 2 or Greater Severity by Day Post Vaccination 3 in Cohort C1 Safety Population

Table 8.2.20 Intestinal Reactogenicity of Grade 2 or Greater Severity by Day Post Any Vaccination in Cohort C1 - Safety Population

| | | Coh | ort C1 | |
|---|---|---|---|---|
| | WRSS1<br>(3 x 10 <sup>3</sup> CFU)<br>(N=XX) | | Pla | cebo<br>I=X) |
| | x/n (%) | 95% CI | x/n (%) | 95% CI |
| Maximum Overall | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Abdominal Pain | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Nausea | | | 1 | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Vomiting | | | 1 | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Loose Stool | | | 1 | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Diarrhoea | • | | • | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| | 1 | | 1 | |

Table 8.2.20 Intestinal Reactogenicity of Grade 2 or Greater Severity by Day Post Any Vaccination in Cohort C1 - Safety Population (continued)

| <b>Dysentery</b> Day 0 Day 1 | (3 x 1 | RSS1<br>03 CFU)<br>=XX)<br>95% CI | | cebo<br>=X) |
|---|---|---|---|---|
| Day 0 | x/n (%) | 95% CI | x/n (%) | |
| Day 0 | | | 7011 (70) | 95% CI |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Bloating | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Excess Flatulence | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |
| Constipation | | | | |
| Day 0 | | | | |
| Day 1 | | | | |
| Day 2 | | | | |
| Day 3 | | | | |

CI = Exact 95% Confidence Interval for the proportion.

- Table 8.2.21 Intestinal Reactogenicity of Grade 2 or Greater by Day Post Vaccination 1 in Cohort C1 - Safety Population
- Table 8.2.22 Intestinal Reactogenicity of Grade 2 or Greater by Day Post Vaccination 2 in Cohort C1 - Safety Population
- Table 8.2.23 Intestinal Reactogenicity of Grade 2 or Greater by Day Post Vaccination 3 in Cohort C1 - Safety Population

Table 8.2.24 Maximum Severity per Participant of Unsolicited Adverse Events Occurring within 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC and PT - Safety Population

| | Cohort C1 | | | |
|---|---|---|---|---|
| | (3 x 1 | RSS1<br>03 CFU)<br>=XX) | | cebo<br>=X) |
| | x/n (%) | 95% CI | x/n (%) | 95% CI |
| Any SOC | | | | |
| Any PT | | | | |
| Mild | | | | |
| Moderate | | | | |
| Severe | | | | |
| Potential Life Threatening | | | | |
| Any Severity | | | | |
| SOC: Specify | <u>. </u> | | <u>. </u> | |
| Any PT | | | | |
| Mild | | | | |
| Moderate | | | | |
| Severe | | | | |
| Potential Life Threatening | | | | |
| Any Severity | | | | |
| SOC: Specify | | | | |
| PT: Specify | | | | |
| Mild | | | | |
| Moderate | | | | |
| Severe | | | | |
| Potential Life Threatening | | | | |
| Any Severity | | | | |

N=Number of participants in the Safety Population.

Cells show frequency (x) and percent of participants with events. n represent number of participants that received vaccination.

CI = Exact 95% Confidence Interval for the proportion.

Note: Table will be extended for other SOC and PT.

- Table 8.2.25 Maximum Severity per Participant of Unsolicited Adverse Events Related to Study Product Occurring Within 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC and PT - Safety Population
- Table 8.2.26 Maximum Severity per Participant of Unsolicited Serious Adverse Events(SAE) Occurring Within 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC and PT Safety Population
- Table 8.2.27 Maximum Severity per Participant of Unsolicited Serious Adverse Events(SAE) Related to Study Product Occurring Within 28 Days After Any Vaccination in Cohort C1, by MedDRA SOC and PT Safety Population
- Table 8.2.28 Maximum Severity per Participant of Unsolicited Adverse Events
  Occurring Within 28 Days After Vaccination 1 in Cohort C1, by
  MedDRA SOC and PT Safety Population
- Table 8.2.29 Maximum Severity per Participant of Unsolicited Adverse Events
  Occurring Within 28 Days After Vaccination 2 in Cohort C1, by
  MedDRA SOC and PT Safety Population
- Table 8.2.30 Maximum Severity per Participant of Unsolicited Adverse Events
  Occurring Within 28 Days After Vaccination 3 in Cohort C1, by
  MedDRA SOC and PT Safety Population
- Table 8.2.31 Maximum Severity per Participant of Unsolicited Adverse Events
  Related to Study Product Occurring Within 28 Days After Vaccination
  1 in Cohort C1, by MedDRA SOC and PT Safety Population
- Table 8.2.32 Maximum Severity per Participant of Unsolicited Adverse Events
  Related to Study Product Occurring Within 28 Days After Vaccination
  2 in Cohort C1, by MedDRA SOC and PT Safety Population
- Table 8.2.33 Maximum Severity per Participant of Unsolicited Adverse Events
  Related to Study Product Occurring Within 28 Days After Vaccination
  3 in Cohort C1, by MedDRA SOC and PT Safety Population

Table 8.2.34 Overall Incidence of Unsolicited Serious Adverse Events Within 28 Days After Vaccination, by Vaccination in Cohort C1 - Safety Population

| | | | Coho | ort C1 | | |
|---|---|---|---|---|---|---|
| | WR:<br>(3 x 10<br>(N= | <sup>3</sup> CFU) | | cebo<br>=X) | | otal<br>=X) |
| | x/n (%) | 95% CI | x/n (%) | 95% CI | x/n (%) | 95% CI |
| Maximum Severity -After Any | Vaccinatio | n | | | | |
| Mild | | | | | | |
| Moderate | | | | | | |
| Severe | | | | | | |
| Potential Life Threatening | | | | | | |
| Any Severity | | | | | | |
| Maximum Severity- After Vac | cination 1 | 1 | • | • | | • |
| Mild | | | | | | |
| Moderate | | | | | | |
| Severe | | | | | | |
| Potential Life Threatening | | | | | | |
| Maximum Severity- After Vac | cination 2 | | | | | |
| Mild | | | | | | |
| Moderate | | | | | | |
| Severe | | | | | | |
| Potential Life Threatening | | | | | | |
| Any Severity | | | | | | |
| Maximum Severity- After Vac | cination 3 | 1 | | | 1 | ı |
| Mild | | | | | | |
| Moderate | | | | | | |
| Severe | | | | | | |
| Potential Life Threatening | | | | | | |
| Any Severity | | | | | | |

Severity is the maximum per participant over all unsolicited adverse events

N=Number of participants in the Safety Population.

Cells show frequency (x) and percent of participants with events. n represent number of participants that received vaccination.

CI = Exact 95% Confidence Interval for the proportion.

Table 8.3.1 Listing of Unsolicited Non-Serious Adverse Events of Grade 2 or Greater Severity in Participants in Cohort C1 - Safety Population

| Adverse<br>Event<br>Description | Onset/<br>End Date | After which vaccination | Onset Day Post- Vaccination | Duration<br>(days) | Severity | Action Taken | Outcome | Relationship<br>to Study<br>Product | MedDRA©<br>System<br>Organ Class | MedDRA©<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Participant xxx | Participant xxxx, WRSS1(3 x 10 <sup>3</sup> CFU) | | | | | | | | | |
| EPIGASTRIC<br>PAIN | 07OCT13 -<br>08OCT13 | 1 | 43 | 2 | Grade 2 | Concomitant<br>Medication | Recovered/ resolved without sequelae | No | Gastrointestinal disorders | Abdominal pain upper |
| Participant yyy | y, Placebo | | | | | | | | | |
| Participant zzzz | z, WRSS1 (3 | x 10 <sup>3</sup> CFU) | | | | | | | | |
| Participant kkk | k, WRSS1 (3 | x 10 <sup>3</sup> CFU) | | | | | | | | |

Table 8.3.2 Listing of Unsolicited Serious Adverse Events in Participants in Cohort C1 - Safety Population

# Table 8.4.1 Listing of all Hematology and Biochemistry Results in Participants in Cohort C1 with any Grade 2 or Greater Severity - Safety Population

Green=Outside the Reference Range, Yellow=Grade 1, Orange=Grade 2, Red=Grade 3, Purple=Grade 4

| | | | | | | | | HEI | MATOL | OGY | | | | | | | | BIO | CHEMIST | RY | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | WBC | Hemo<br>globin | Plate<br>lets | Neutr | rophils | Lymph | nocytes | Mono | cytes* | Eosin | ophils | Baso | phils* | ESR* | RBC* | Creat inine | AST | ALT<br>(SGPT) | GGT | Total<br>Bili<br>rubin |
| Visit | Age<br>(Years) | 10 <sup>9</sup> /L | gm/dL | 10 <sup>9</sup> /L | % | cells/<br>mm <sup>3</sup> | % | cells/<br>mm³ | % | 10 <sup>9</sup> /L | % | 10 <sup>9</sup> /L | % | 10 <sup>9</sup> /L | m/<br>1 <sup>st</sup> hr | 10 <sup>12</sup> /L | U/L | umol/<br>L | U/L | | umol/<br>L |
| Particip | ant 11012 | , WRS | S1 (3 x 10 | <sup>4</sup> CFU) | • | | | | | | • | | | • | • | • | • | • | | | |
| Screen<br>-ing | | | | | | | | | | | | | | | | | | | | | |
| Day 7 | | | | | | | | | | | | | | | | | | | | | |
| Particip | ipant 11019, WRSS1 (3 x 10 <sup>5</sup> CFU) | | | | | | | | | | | | | | | | | | | | |
| Screen<br>-ing | | | | | | | | | | | | | | | | | | | | | |
| Day 7 | | | | | | | | | | | | | | | | | | | | | |
| Particip | ant 11042 | , WRS | S1 (3 x 10 | <sup>5</sup> CFU) | | | | | | | | | | | | | | | | | |
| Screen<br>-ing | | | | | | | | | | | | | | | | | | | | | |
| Day 7 | | | | | | | | | | | | | | | | | | | | | |
| Particip | icipant 11050, Placebo | | | | | | | | | | | | | | | | | | | | |
| Screen<br>-ing | | | | | | | | | | | | | | | | | | | | | |
| Day 7 | | | | | | | | | | | | | | | | | | | | | |

# Table 8.5.1 Listing of all Physical Examination and Vital Signs Values in Participants in Cohort C1 with Any Abnormality Findings - Safety Population

Yellow=Abnormal NCS, Red=Abnormal, CS

| | | | | | | Physica | I Examination | 1 | | | | Vi | tal Sign | S | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Cardio- | | | Musculo- | | Heart<br>Rate | Respi<br>Ra | ratory<br>ite | Axi<br>Temp | llary<br>erature |
| Visit | Age<br>(Years) | HEENT | Skin | Lymph<br>Nodes | Respiratory<br>(Lung) | | Abdomen | Neurological | skeletal<br>System | Other | Beats/<br>minute | Breaths/<br>minute | | °C | |
| Participa | ant 11012, | 12, WRSS1 (3 x 10⁴ CFU) | | | | | | | | | | | | | |
| Screeni<br>ng | | | | | | | | | | | | | | | |
| Day 7 | | | | | | | | | | | | | | | |
| Day 28 | | | | | | | | | | | | | | | |
| Day 35 | | | | | | | | | | | | | | | |
| Day 56 | | | | | | | | | | | | | | | |
| Day 63 | | | | | | | | | | | | | | | |
| Day 84 | | | | | | | | | | | | | | | |
| Participa | ant 11019, | WRSS1 ( | 3 x 10 <sup>5</sup> C | FU) | | | | | | | | | | | |
| Screeni<br>ng | | | | | | | | | | | | | | | |
| Day 7 | | | | | | | | | | | | | | | |
| Day 28 | | | | | | | | | | | | | | | |
| Day 35 | | | | | | | | | | | | | | | |
| Day 56 | | | | | | | | | | | | | | | |
| Day 63 | | | | | | | _ | | | | | | | | |
| Day 84 | | | | | | | | | | | | | | | |

Table 10.2.1 IgA Antibodies in ALS, Descriptive Statistics - Per Protocol Population

| | Inv | aplex | I | LPS |
|---|---|---|---|---|
| | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) |
| Day 0 | | | | <u> </u> |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |
| Day 7 | | | | |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |
| Day 35 | | | | <u> </u> |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |
| Day 63 | | | | , |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |

N=Number of participants in the Per-Protocol Population and n=Number of participants with non-missing values. SD = Standard Deviation. GMT = Geometric Mean titer.

Table 10.2.2 IgG Antibodies in ALS, Descriptive Statistics - Per Protocol Population Table 10.2.3 IgM Antibodies in ALS, Descriptive Statistics - Per Protocol Population Same as 10.2.1

Table 10.2.4 Fold-Rise from Baseline in IgA Antibodies in ALS – Per-Protocol Population

| | Inv | aplex | L | PS |
|---|---|---|---|---|
| | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) |
| Day 7 | | | | |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |
| Ratio (95% CI) <sup>1</sup> | | | | |
| Day 35 | | | | |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |
| Ratio (95% CI) <sup>1</sup> | | | | |
| Day 63 | | | | |
| n | | | | |
| Mean (SD) Log titer | | | | |
| GMT | | | | |
| 95% CI for GMT | | | | |
| Median | | | | |
| Range | | | | |
| Ratio (95% CI) <sup>1</sup> | | | | |

N=Number of participants in the Per-Protocol Population and n=Number of participants with non-missing values SD = Standard Deviation. GMT = Geometric Mean titer.

Table 10.2.5 Fold-Rise from Baseline in IgG Antibodies in ALS – Per-Protocol Population

Table 10.2.6 Fold-Rise from Baseline in IgM Antibodies in ALS – Per-Protocol Population

Same as 10.2.4

<sup>&</sup>lt;sup>1</sup> WRSS1 versus Placebo ratio, back-transformed estimates from Student's Test of difference between mean Log Titers.

# Table 10.2.7 4-Fold Rise<sup>1</sup> in IgA Antibodies in ALS Proportion of Participants with at Least a 4-Fold Rise from Baseline – Per-Protocol Population

| | Inv | /aplex | | LPS |
|---|---|---|---|---|
| | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) |
| Day 7 | | | | |
| Number of observations | | | | |
| n (%) | | | | |
| 95% CI | | | | |
| P-Value <sup>2</sup> | 0 | .xxxx | 0 | .xxxx |
| Day 35 | | <u> </u> | | |
| Number of observations | | | | |
| n (%) | | | | |
| 95% CI | | | | |
| P-Value <sup>2</sup> | 0 | .xxxx | 0 | .xxxx |
| Day 63 | | - | | |
| Number of observations | | | | |
| n (%) | | | | |
| 95% CI | | | | |
| P-Value <sup>2</sup> | 0 | .xxxx | 0 | .xxxx |
| At Any Time | | | | |
| Number of observations | | | | |
| n (%) | | | | |
| 95% CI | | | | |
| P-Value <sup>2</sup> | 0 | .xxxx | 0.xxxx | |

N=Number of participants in the Per-Protocol Population and n=Number of participants with non-missing values CI = Exact (Clopper-Pearson) Confidence Interval for the proportion.

<sup>&</sup>lt;sup>1</sup> Fold rise is the ratio of follow-up titer/baseline titer. For those with a zero titer on Day 1, fold-rise was defined as the follow-up titer.

<sup>&</sup>lt;sup>2</sup> Fisher's exact 2-tailed test of a difference in proportions between WRSS1 and Placebo.

- Table 10.2.8 4-Fold Rise in IgG Antibodies in ALS Proportion of Participants with at Least a 4-Fold Rise from Baseline Per-Protocol Population
- Table 10.2.9 4-Fold Rise in IgM Antibodies in ALS Proportion of Participants with at Least a 4-Fold Rise from Baseline Per-Protocol Population
- Table 10.2.10 Table 10.2.12 Replicate Table 10.2.1-10.2.3 for IgA, IgG and IgM Antibodies in Serum
- Table 10.2.13 Table 10.2.15 Replicate Table 10.2.4-10.2.6 for IgA, IgG and IgM Antibodies in Serum
- Table 10.2.16 Table 10.2.18 Replicate Table 10.2.7-10.2.9 for IgA, IgG and IgM Antibodies in Serum
- Table 10.2.19 Replicate Table 10.2.1 for IgA Antibodies in Stool Per Protocol Population, include extra visits (Days 28, 56 and 84)
- Table 10.2.20 Replicate Table 10.2.4 for IgA Antibodies in Stool Per Protocol Population, include extra visits (Days 28, 56 and 84)
- Table 10.2.21 Replicate Table 10.2.7 for IgA Antibodies in Stool Per Protocol Population, include extra visits (Days 28, 56 and 84)

Table 10.2.22 Proportion of Participants with WRSS1 Shedding at Any Time after Vaccination – Per-Protocol Population

| | Placebo<br>(N=XX) | WRSS1 3x10 <sup>3</sup><br>(N=XX) |
|---------|-------------------|-----------------------------------|
| N. Obs. | Х | xx |
| n (%) | x (xx.x) | x (xx.x) |
| 95% CI | (0.xx - xx.x) | (0.xx – xx.x) |

N=Number of participants in the Per-Protocol Population and n=Number of participants with non-missing values

Fisher's exact 2-tailed test of a difference in proportions between WRSS1 and Placebo: p=0.xxxx

N. Obs.= Number of observations

CI = exact confidence interval

#### **Other Listings**

- 1. Listing of Participants Withdrawn
- 2. Listing of Demographic and Other Baseline Characteristics
- 3. Listing of Medical History
- 4. Listing of Physical Examination Results
- 5. Listing of Protocol Deviations
- 6. Listing of Participant Vaccinations